CLINICAL TRIAL: NCT03970239
Title: Role of the Serotoninergic System in Impulse Control Disorders in Parkinson's Disease
Brief Title: Serotonin in Impulse Control Disorders in Parkinson's Disease
Acronym: Park-IMPULSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL18_0012; 2019-000340-99 (EudraCT Number)
Record Dates: First submitted 2019-05-06; First posted 2019-05-31 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-02

CONDITIONS: Parkinson Disease; Impulse Control Disorders
Keywords: Parkinson's disease; Impulse control disorders; Serotoninergic system; Positron Emission Tomography (PET)
MeSH Terms: conditions — Parkinson Disease; Disruptive, Impulse Control, and Conduct Disorders | interventions — 3-amino-4-(2-dimethylaminomethylphenylsulfanyl)benzonitrile

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson's Disease patients (Experimental): All study participants undergo functional imaging of the serotoninergic system with Positron Emission Tomography (PET) using [11 Carbon]-3-amino-4-(2-dimethylaminomethylphenylsulfanyl)-benzonitrile ([11C]-DASB) and [18 Fluorine]-altanserin ([18F]-altanserin). [11C] -DASB is a highly specific PET radiotracer which binds to the serotonin transporter (SERT).
  [18F]-altanserin is a highly specific PET radiotracer which specifically binds to the serotonin 5-hydroxytryptamine receptor 2A (5-HT2A) receptor.
  Interventions: Drug: Positron Emission Tomography using [11 Carbon]-3-amino-4-(2-dimethylaminomethylphenylsulfanyl)-benzonitrile ([11C]-DASB) and [18 Fluorine]-altanserin ([18F]-altanserin)
- Imaging of healthy volunteers (Experimental): All healthy volunteers undergo functional imaging of the serotoninergic system with Positron Emission Tomography (PET) using [18F]-altanserin.
  [18F]-altanserin is a highly specific PET radiotracer which specifically binds to the serotonin 5-hydroxytryptamine receptor 2A (5-HT2A) receptor.
  Interventions: Drug: Positron Emission Tomography using [18 Fluorine]-altanserin ([18F]-altanserin)

INTERVENTIONS:
Drug: Positron Emission Tomography using [11 Carbon]-3-amino-4-(2-dimethylaminomethylphenylsulfanyl)-benzonitrile ([11C]-DASB) and [18 Fluorine]-altanserin ([18F]-altanserin) — Imaging of the serotoninergic system with Positron Emission Tomography using [11 Carbon]-3-amino-4-(2-dimethylaminomethylphenylsulfanyl)-benzonitrile ([11C]-DASB) and [18 Fluorine]-altanserin ([18F]-altanserin). During this study, subjects will receive a single intravenous administration of approximately 4 Megabecquerel/kilogram (MBq/kg) of [11C]-DASB immediately prior to imaging using Positron Emission Tomography (PET). The effective dose in human body is about 2.1 milliSievert (mSv).
  On a separate day, subjects will receive a single intravenous administration of approximately 3.7 MBq/kg of [18F]-altanserin for 120 minutes prior to imaging using Positron Emission Tomography (PET). The effective dose in human body is about 8.4 mSv.
  Arms: Parkinson's Disease patients
Drug: Positron Emission Tomography using [18 Fluorine]-altanserin ([18F]-altanserin) — Imaging of the serotoninergic system with Positron Emission Tomography using [18 Fluorine]-altanserin ([18F]-altanserin). During this study, subjects will receive a single intravenous administration of approximately 3.7 Megabecquerel/kilogram (MBq/kg) of [18F]-altanserin 120 minutes prior to imaging using Positron Emission Tomography. The effective dose in human body is about 8.4 mSv.
  Arms: Imaging of healthy volunteers

SUMMARY:
Impulse control disorders are frequent and troublesome in patients with Parkinson's disease. However, the cerebral functional alterations related to impulse control disorders in Parkinson's disease are poorly understood and may involve the serotoninergic system besides alterations in the dopaminergic system.

The primary objective of this study is to investigate the cerebral functional alterations in the serotoninergic system in patients with Parkinson's disease and impulse control disorders using Positron Emission Tomography with highly specific radiotracers of serotonin transporter (SERT) using [11 Carbon]-3-amino-4-(2-dimethylaminomethylphenylsulfanyl)-benzonitrile ([11C]-DASB) and of serotonin 5-Hydroxytryptamine 2A (5-HT2A) receptor using [18 Fluorine]-altanserin ([18F]-altanserin), in comparison to patients with Parkinson's disease without impulse control disorders and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Group 1 Patients with Parkinson's disease and impulse control disorders

* Patients with a diagnosis of clinically established or clinically probable Parkinson's disease according to the Movement Disorder Society (MDS) Clinical Diagnostic Criteria for Parkinson's Disease
* Patients aged ≥ 30 and ≤ 80 years old
* Patients presenting currently with impulse control disorders or having presented with impulse control disorders in the last 2 years (Ardouin Behavior Scale score ≥2 for one or more of the following items: eating behavior; compulsive buying; pathological gambling; hypersexuality) , following the diagnosis of Parkinson's disease
* Patients able to sign the consent document and willing to participate in all aspects of the study

Patients with Parkinson's disease and without impulse control disorders

* Patients with a diagnosis of clinically established or clinically probable Parkinson's disease according to the MDS Clinical Diagnostic Criteria for Parkinson's Disease
* Patients aged ≥ 30 and ≤ 80 years old
* Patients not currently presenting with impulse control disorders and other hyperdopaminergic behaviors and not having ever presented with impulse control disorders
* Patients able to sign a consent document and willing to participate in all aspects of the study

Group 2 : Healthy volunteers

Subjects aged ≥ 30 and ≤ 80 years old

* Subjects not currently presenting with impulse control disorders or hyperdopaminergic behaviors and not having ever presented with impulse control disorders
* Subjects able to sign a consent document and willing to participate in all aspects of the study

Exclusion Criteria:

Group 1 :

Patients with Parkinson's disease and impulse control disorders

* Patients with Montreal Cognitive Assessment score ≤24 or Frontal Assessment Battery score ≤14
* Patients not able to perform Positron Emission Tomography (PET) or Magnetic Resonance Imaging (MRI)
* Patients presenting with other severe medical condition or other parkinsonian syndrome
* Patients treated with Deep Brain Stimulation or levodopa pump
* Patients treated with drugs or consuming recreative drugs specifically interfering with the serotoninergic, noradrenergic or opiate systems in the last 3 months
* Patients presenting with substance dependence, except for tobacco
* Patients with Body Mass Index ≥ 35kilogram/meters2 (kg/m2)

Patients with Parkinson's disease and without impulse control disorders

* Patients with Montreal Cognitive Assessment score ≤24 or Frontal Assessment Battery score ≤14
* Patients not able to perform Positron Emission Tomography or Magnetic Resonance Imaging
* Patients presenting with other severe medical condition or other parkinsonian syndrome
* Patients treated with Deep Brain Stimulationor levodopa pump
* Patients treated with drugs or consuming recreative drugs specifically interfering with the serotoninergic, noradrenergic or opiate systems in the last 3 months
* Patients presenting with substance dependence, except for tobacco
* Patients with Body Mass Index ≥35kg/m2

Group 2 : Healthy volunteers

* Subjects with Montreal Cognitive Assessment score ≤24 or Frontal Assessment Battery score ≤14
* Subjects not able to perform Positron Emission Tomography or Magnetic Resonance Imaging
* Subjects presenting with neurologic, psychiatric or other severe medical condition
* Subjects treated with drugs or consuming recreative drugs specifically interfering with the serotoninergic, noradrenergic or opiate systems in the last 3 months
* Subjects presenting with substance dependence, except for tobacco
* Subjects with Body Mass Index ≥35kg/m2

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-05-13 (Actual); Primary Completion 2022-02-13 (Estimated); Study Completion 2022-02-13 (Estimated)

PRIMARY OUTCOMES:
Difference in binding potential of [18 Fluorine]-altanserin ([18F]-altanserin) and [11 Carbon]-3-amino-4-(2-dimethylaminomethylphenylsulfanyl)-benzonitrile ([11C]-DASB) ([11C]-DASB) | 2-3 days
  Between-group difference of binding potential of [18 Fluorine]-altanserin ([18F]-altanserin) and [11 Carbon]-3-amino-4-(2-dimethylaminomethylphenylsulfanyl)-benzonitrile ([11C]-DASB) ([11C]-DASB)

SECONDARY OUTCOMES:
Ardouin Scale of Behavior in Parkinson's Disease (ASBPD) | 2-3 days
  The Ardouin Scale of Behavior in Parkinson's Disease (ASBPD) evaluates hypo- and hyperdopaminergic behaviors and can also detect and quantify neuropsychiatric fluctuations by evaluating OFF-drug dysphoria and ON-drug euphoria. It is based on a semi-structured interview that encompasses the whole spectrum of behavioral spectrum from hypo-to hyperdopaminergic syndromes as well as non-motor fluctuations. The scale consists of 18 items addressing non-motor symptoms, grouped in four parts: general psychological evaluation, apathy, non-motor fluctuations and hyperdopaminergic behaviors. The rating in five points (0-4 from absent to severe) is carried out during a semi-structured interview. Open-ended questions introduce each item, allowing patients to express themselves as freely as possible. Close-ended questions permit the rating of severity and intensity.
Questionnaire For Impulsive-Compulsive Disorders In Parkinson's Disease-Rating Scale (QUIP-RS) | 2-3 days
  The Questionnaire For Impulsive-Compulsive Disorders In Parkinson's Disease-Rating Scale (QUIP-RS) is designed to measure severity of symptoms and support a diagnosis of impulse control disorders and related disorders in Parkinson's Disease (PD). The QUIP-RS is administered with an instruction sheet that provides examples of the behaviors being assessed and a brief description of the categories for frequency (never [0] = not at all, rarely [1] = infrequently or 1 day/week, etc.). Scores for each Impulsive Compulsive Disorder (ICD) and related disorder range from 0 to 16, with a higher score indicating greater severity (frequency) of symptoms. The total QUIP-RS score for all ICDs and related disorders combined ranges from 0 to 112.
Urgency, Premeditation (lack of), Perseverance (lack of), Sensation Seeking Impulsive Behavior Scale (UPPS Impulsive Behavior Scale) | 2-3 days
  The full version of the UPPS-P Scale is composed of 59 items, with 10-14 items per scale. Items are scored on a 4-point scale:
  Agree Strongly = 1 Agree Some = 2 Disagree Some = 3 Disagree Strongly = 4
  Higher values translate into higher levels of impulsivity. The results allow assessement of the patient according to five impulsive personality traits:
  * Negative urgency: tendency to act rashly under extreme negative emotions
  * Lack of Premeditation: tendency to act without thinking
  * Lack of Perseverance: inability to remain focused on a task
  * Sensation Seeking: tendency to seek out novel and thrilling experiences
  * Positive Urgency: tendency to act rashly under extreme positive emotions
Movement Disorder Society (MDS) Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 2-3 days
  The MDS-UPDRS is composed of four parts, namely, I: Non-motor Experiences of Daily Living; II: Motor Experiences of Daily Living; III: Motor Examination; IV: Motor Complications and includes 65 items. Each question has five responses that are linked to commonly accepted clinical terms: 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The overall progression of disability is given a score ranging from 0 = no disability 1= slight disability 2= moderate disability 3= high disability and 4= severe disability.
Beck Depression Inventory II (BDI-II) | 2-3 days
  The Beck Depression Inventory (BDI-II) is used to measure the severity of depression. It contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms:
  * 0-13: minimal depression
  * 14-19: mild depression
  * 20-28: moderate depression
  * 29-63: severe depression.
Starkstein Apathy Scale (SAS) | 2-3 days
  For this scale, patients are asked to answer 14 questions, each of which is scored on a 4-point scale of 0-3, and apathy is rated as more severe as the total score (0-42) increases.
State-Trait Anxiety Inventory -Y (STAI-Y) | 2-3 days
  The State-Trait Anxiety Inventory measures anxiety by assessing someone's state (S) and trait (T) anxiety at the same time. Its combined format consists of 40 questions. The S-Anxiety scale (STAI Form Y-1) consists of twenty statements that evaluate how the respondent feels "right now, at this moment". The T- Anxiety scale (STAI Form Y-2) consists of twenty statements that evaluate how the respondent feels "generally". In responding to the S-Anxiety scale, the subjects choose the number that best describes the intensity of their feelings: (1) not at all, (2) somewhat, (3) moderately, (4) very much so. In responding to the T-Anxiety scale, subjects rate the frequency of their feelings on the following four-point scale: (1) almost never, (2) sometimes, (3) often, (4) almost always. Each STAI item is given a weighted score of 1 to 4. Scores for both the S-Anxiety and the T-Anxiety scales can vary from a minimum of 20 to a maximum of 80 with higher scores correlating to higher anxiety.
Snaith-Hamilton Pleasure Scale (SHAPS) | 2-3 days
  The SHAPS measures the subject's ability to experience pleasure (hedonic tone) and its absence (anhedonia). It consists of 14 items with 4 possible responses: Definitely Agree, Agree, Disagree, Definitely Disagree. A score from 0- 14 is possible (1 point for each response in the Disagree category and 0 points for each response in the Agree category). The higher the score the less the subject is able to experience pleasure.
Temporal Experience of Pleasure Scale (TEPS) | 2-3 days
  Measure specifically designed to capture the anticipatory and consummatory facets of pleasure. It consists of 10 questions assessing anticipatory pleasure (TEPS-ANT) and 8 questions assessing consummatory pleasure (TEPS-CON) using a 6-point fixed choice response format ranging from 1 = very false for me to 6 = very true for me. The higher the score for each section, the more the subject experiences anticipatory pleasure and consummatory pleasure, respectively.
Stop Signal Reaction Time (SSRT) | 2-3 days
  Stop Signal Task
Discounting rate | 2-3 days
  27-item Monetary Choice Questionnaire: for each question, patients will choose between two different monetary values (a high monitary value versus a low monitary value) in order to determine the patient's level of impulsiveness.
Proportion of premature responses | 2-3 days
  4 Choice Serial Reaction Time Task
Polymorphism rs6313 (or T102C) of the serotonin 5-Hydroxytryptamine 2A (5-HT2A) receptor | 2-3 days
  Polymorphism rs6313 also called T102C or C102T is a gene variation, a single nucleotide polymorphism (SNP) in the human Hydroxytryptamine Receptor 2A (HTR2A) gene that codes for the 5-HT2A receptor. The SNP is a synonymous substitution located in exon 1 of the gene where it is involved in coding the 34th amino acid as serine.
Polymorphism 5-HydroxyTryptamine (serotonin) Transporter Gene-Linked Polymorphic Region (5-HTTLPR)/rs25531 of the serotonin transporter (SERT) | 2-3 days
  Polymorphism 5-HydroxyTryptamine (serotonin) Transporter Gene-Linked Polymorphic Region (5-HTTLPR)/rs25531 of the serotonin transporter (SERT)
Magnetic Resonance Imaging metrics: anatomical imaging | 2-3 days
  Anatomical imaging using a T1-weighted Magnetization-Prepared RApid Gradient-Echo (T1_MPRAGE) sequence for morphometry.
Magnetic Resonance Imaging metrics: Diffusion Weighted imaging | 2-3 days
  Diffusion weighted imaging for Diffusion Tensor Imaging (DTI) and tractography
Magnetic Resonance Imaging metrics: Resting State Functional Imaging | 2-3 days
  Resting State Functional Imaging for functional connectivity

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane THOBOIS, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France